CLINICAL TRIAL: NCT02834754
Title: A Randomized, Double-blind, Placebo Controlled Study of Vedolizumab for the Prevention of Post-operative Crohn's Disease Recurrence
Brief Title: Vedolizumab Post Op Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited time for enrollment of required number of subjects
Sponsor: Marc Schwartz (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Marc Schwartz, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO16030443
Record Dates: First submitted 2016-07-12; First posted 2016-07-15 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Crohn's Disease
Keywords: post-operative
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vedolizumab (Experimental): Vedolizumab infusions at weeks 0, 2, and 6 weeks, then every 8 weeks for 52 weeks
  Interventions: Drug: Vedolizumab
- placebo (Placebo Comparator): Placebo infusions at weeks 0, 2, and 6 weeks, then every 8 weeks for 52 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab is a monoclonal antibody developed by Millennium Pharmaceuticals, Inc for the treatment of ulcerative colitis and Crohn's disease. It binds to integrin α₄β₇. Blocking the α₄β₇ integrin results in gut-selective anti-inflammatory activity. Vedolizumab was been approved by the Food and Drug Administration (FDA) in 2014 for achieving clinical response, achieving clinical remission, and achieving corticosteroid-free remission in adult patients with moderately to severely active Crohn's disease. We believe that use of vedolizumab constitutes a non-significant risk to the research subject. The dose of vedolizumab administered is 300mg IV
  Other Names: entyvio
  Arms: Vedolizumab
Drug: placebo — Currently there are no clinical guidelines and no standard of care for the maintenance of surgically induced remission. There are no medications that have consistently been proven to be efficacious at preventing recurrent Crohn's disease and as such, no active equivalent arm is being used. Due to the lack of effective prophylactic therapy, many physicians and patients opt not to initiate medical therapy after surgery, rather wait until Crohn's disease recurs, or wait to perform a post-operative colonoscopy within 6-12 months of surgery, and decide on initiating Crohn's disease therapy based on endoscopic Rutgeerts; score. Therefore, acknowledging that many patients are not administered post-operative maintenance medications, we feel the placebo arm is justified.
  Arms: placebo

SUMMARY:
This is a pilot study that will determine the endoscopic recurrence of Crohn's disease 12 months after curative, resective ileal or ileocolonic surgery in patients receiving post-operative vedolizumab (Entyvio) or placebo. The investigators hypothesize that the administration of post-operative vedolizumab will decrease the endoscopic recurrence of Crohn's disease.

DETAILED DESCRIPTION:
Study aims: To determine the efficacy of vedolizumab in preventing mucosal recurrence of Crohn's disease in patients undergoing resective surgery.

Methods: This is a randomized, placebo-controlled pilot study that will determine the endoscopic recurrence of Crohn's disease 12 months after curative, resective ileal or ileocolonic surgery in patients receiving post-operative vedolizumab or placebo. Patients will receive the first infusion of vedolizumab (300 mg) or placebo (1:1 randomization) 2-4 weeks after surgery. Subsequent infusions of vedolizumab or placebo will occur at 2, 6, 14, 22, 30, 38, 46, and 54 weeks after the first infusion. The primary assessment for determination of drug efficacy will be presence or absence of mucosal inflammation (representing active Crohn's disease) at the ileocolonic anastomosis and neo-terminal ileum. This assessment will be made by colonoscopic inspection one year after surgery. Patients with an elevated fecal calprotectin at week 22 will undergo a 6-month post-operative clinical colonoscopy to assess for endoscopic recurrence.

Subject population: Patients scheduled for resectional surgery for ileal or ileocolonic Crohn's disease will be eligible for the study. Subjects will be male or female who are 18 years of age or older.

ELIGIBILITY:
Inclusion Criteria:

1. Are men or women > 18 years of age at screening.
2. Curative resection and ileocolonic anastomosis for Crohn's disease. Patients with isolated fibrostenotic (non-inflammatory) or minimal (not clinically significant) disease elsewhere in gastrointestinal that is not resected will also be included.
3. Participants who have received pre-operative vedolizumab therapy may be included.
4. Concomitant medications: All concomitant medications at the time of the surgery will be discontinued post-operatively.
5. Men and women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) for the duration of the study and should continue such precautions for 6 months after receiving the last infusion).
6. Antibiotics for the treatment of Crohn's disease (eg. ciprofloxacin and metronidazole) are allowable but must be discontinued within 12 weeks after surgery. Antibiotics for the treatment of a concomitant infection are allowable throughout the duration of the study as long as the primary purpose of antibiotic therapy is not for the primary treatment of Crohn's disease.
7. Screening laboratory tests must meet the screening criteria (Hemoglobin ≥ 8.5 g/dL, White blood cell (WBC) count ≥ 3.0 x 109/L, Neutrophils ≥ 1.0 x 109/L, Platelets ≥ 100 x 109/L, Lymphocyte count ≥ 0.5 x 109/L and SGOT (AST-aspartate aminotransferase) -< 3 times upper normal limit).
8. Are capable of providing written informed consent, and the consent must be obtained prior to conducting any protocol-specified procedures.
9. Are willing to adhere to the study visit schedule and other protocol requirements.
10. Participants who require a temporary diverting ileostomy and then takedown will be included. These would be participants who undergo resective surgery and primary ileocolonic anastomosis but require a temporary diverting ostomy proximal to the anastomotic site. Participants will be eligible for the study upon takedown of the diverting ileostomy

Exclusion Criteria:

1. Participants with greater than 10 years of Crohn's disease requiring their FIRST resection of a short (<10cm) fibrostenotic stricture. The rationale for excluding these participants is that historically this group of participants is at a very low risk of recurrence and therefore, would not be a group targeted for postoperative medical therapy.
2. Macroscopically active disease at the anastomosis at the time of surgery.
3. Presence of a stoma.
4. Prior severe infusion reaction to vedolizumab, i.e. anaphylaxis, bronchospasm, or hypotension.
5. History of anaphylaxis to other chimeric proteins.
6. Any of the following medications taken within 12 weeks of surgery: cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, or other investigational drugs. Patients who have taken these medications more than 12 weeks prior to surgery will be allowed in the study
7. At the time of screening participants with a positive stool culture for enteric pathogens, pathogenic ova or parasites, or Clostridium difficile toxin and have clinically significant signs of an enteric infection, i.e. diarrhea, fever, abdominal pain. participants will be eligible for enrollment if stool cultures are positive but do not have clinically significant signs or symptoms or infection and receive appropriate antibiotic treatment. A repeat stool culture will be obtained at the completion of antibiotic treatment.
8. Women who are pregnant, nursing, or planning pregnancy during the trial or within 6 months after the last infusion (this includes father's who plan on fathering a child within 6 months after their last infusion).
9. Have or have had an opportunistic infection (eg, herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months of screening.
10. Have a chest radiograph within 3 months prior to screening that shows evidence of malignancy, infection, or any abnormalities.
11. Documentation of seropositive for human immunodeficiency virus (HIV).
12. Documentation of a positive test for hepatitis B surface antigen or a history of documented hepatitis C.
13. Have current signs or symptoms of systemic lupus erythematosus, or severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral diseases.
14. Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to randomization).
15. Have any current known malignancy other than the condition being treated or have a history of malignancy within 5 years prior to screening (except for squamous or basal cell carcinoma of the skin that has been fully excised with no evidence of recurrence).
16. Have a history of lymphoproliferative disease including lymphoma, or signs or symptoms suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (eg, nodes in the posterior triangle of the neck, intraclavicular, epitrochlear, or periaortic area), or splenomegaly.
17. Have had a known substance abuse (drug or alcohol) or dependency within the previous 3 years, history of noncompliance to medical regimens, or other condition/circumstance that could interfere with the subject's adherence to protocol requirements (eg, psychiatric disease, lack of motivation, travel, etc).
18. Are unable to or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access
19. Have had a chronic or recurrent infectious disease including, but not limited to, chronic renal infection, chronic chest infection (eg, bronchiectasis), sinusitis, recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), open, draining, or infected skin wound, or ulcer.
20. Have had a serious infection (eg, hepatitis, pneumonia, or pyelonephritis), have been hospitalized for an infection, or have been treated with intravenous (IV) antibiotics for an infection within 2 months prior to randomization. The exception being participants whose infection is a direct consequence of their Crohn's disease and will be completely resolved with surgery, e.g. participants with an abscess related to penetrating Crohn's disease of the terminal ileum who have no sign of infection after surgery. Less serious infections (eg, acute upper respiratory tract infection, enteric infections without signs or symptoms or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator.
21. Have a serious concomitant illness that could interfere with the subject's participation in the trial.
22. Current use of prescription doses or chronic and frequent use of over-the-counter doses of nonsteroidal anti-inflammatory drugs (NSAIDs), except low-dose aspirin for prevention of heart attacks, unstable angina, or transient ischemic attacks.
23. Have ulcerative colitis.
24. Are participating in another investigative trial during participation in this trial.
25. Use of any investigational drug within 30 days prior to randomization or within 5 half-lives of the investigational agent, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Endoscopic remission | 54 weeks
  During a follow up colonoscopy, the Rutgeerts' score will be used to assess for endoscopic remission. An endoscopy score of i0 or i1 will be considered endoscopic remission and a score of i2 or higher denotes endoscopic recurrence. The endoscopic scoring system is as follows: Grade 0 normal distal ileum, Grade 1 up to 5 small aphthous ulcers, Grade 2 six or more aphthous ulcers with skip areas either at the ilocolonic anastomosis or proximal to it, Grade 3 diffuse aphthous ileitis with diffusely inflamed mucosa and Grade 4 diffuse inflammation with larger ulcers, nodules, and/or narrowing.

SECONDARY OUTCOMES:
clinical remission | 54 weeks
  CDAI <150
Histologic remission | 54 weeks
  Geboes score

CONTACTS AND LOCATIONS:
Overall Officials: Marc B Schwartz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States